CLINICAL TRIAL: NCT04296409
Title: The Turkish Version of the Deglutition Handicap Index
Brief Title: The Turkish Deglutition Handicap Index
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, SELEN SEREL ARSLAN, Principal Investigator, Hacettepe University
Other Study IDs: Dysphagia evaluation
Record Dates: First submitted 2020-03-03; First posted 2020-03-05 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Swallowing Disorder
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult patients with swallowing disorders: Swallowing function will be evaluated with the Turkish Deglutition Handicap Index, and Turkish version of the Eating Assessment Tool.
  Interventions: Other: Turkish Deglutition Handicap Index

INTERVENTIONS:
Other: Turkish Deglutition Handicap Index — Swallowing function will be evaluated by the Turkish Deglutition Handicap Index.

SUMMARY:
The purpose of this study is to test the reliability and validity of the The Turkish Deglutition Handicap Index among adult patients with swallowing disorders.

DETAILED DESCRIPTION:
The purpose of this study is to test the reliability and validity of the The Turkish Deglutition Handicap Index among adult patients with swallowing disorders.The internal consistency, test-retest reliability, and criterion validity of the instrument will be investigated. The internal consistency will be assessed using Cronbach's alpha. Intraclass correlation coefficient (ICC) value with 95 % confidence intervals will be calculated for test-retest reliability. The criterion validity of the scale will be determined by assessing the correlation between The Turkish Deglutition Handicap Index and Turkish Eating Assessment Tool.

ELIGIBILITY:
Inclusion Criteria:

* Willing to participate
* Having swallowing problems

Exclusion Criteria:

* Being under the age of 20 years, and above the age of 60 years
* Not willing to participate
* Having no swallowing problems

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Adult patients with swallowing difficulties
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2022-06-22 (Actual); Primary Completion 2023-02-22 (Actual); Study Completion 2023-02-22 (Actual)

PRIMARY OUTCOMES:
Turkish Deglutition Handicap Index | 3 months
  Turkish Deglutition Handicap Index is a swallowing function evaluation tool. The test consists of 30 items which will be scored between 0 to 4. 0 means Never, and 4 means Always. The test score ranges from 30 (minimum) to 120 (maximum) points.

SECONDARY OUTCOMES:
The Turkish version of the Eating Assessment Tool-10 | 3 months
  The Turkish version of the Eating Assessment Tool-10 is a self-reporting instrument with 10 questions. Total score ranges between 0 to 40. Higher scores indicate worse swallowing function.

CONTACTS AND LOCATIONS:
Overall Officials: SELEN SEREL ARSLAN, Principal Investigator — Hacettepe University
Locations (1):
- Hacetttepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No